CLINICAL TRIAL: NCT00357630
Title: Phase II Protocol: Gemcitabine for Metastatic Cancer With Unknown Primary Site - Analysis of Symptom Benefit
Brief Title: Gemcitabine in Treating Patients With Metastatic Cancer of Unknown Primary
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert L. Comis, ECOG Group Chair's Office
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000486704; ECOG-E5Z02
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2008-10

CONDITIONS: Carcinoma of Unknown Primary; Pain
Keywords: adenocarcinoma of unknown primary; newly diagnosed carcinoma of unknown primary; undifferentiated carcinoma of unknown primary; pain
MeSH Terms: conditions — Neoplasms, Unknown Primary; Pain | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well gemcitabine works in treating patients with metastatic cancer of unknown primary.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of gemcitabine hydrochloride in patients with metastatic cancer of unknown primary (CUP), in terms of improved quality of life (QOL) (as measured by the FACT Physical Well Being subscale [FACT-G]) and reduction of symptom distress (as measured by the Memorial Symptom Assessment Scale Short Form Global Distress Index [MSAS-SF]).
* Define clinical benefit response using a QOL instrument in patients with CUP receiving gemcitabine hydrochloride.
* Correlate objective and/or evaluable tumor response with symptom and QOL response in these patients.
* Explore the association between symptom response, QOL response, and clinical benefit response in these patients.
* Evaluate changes in QOL in patients who have no symptom or objective response after treatment with gemcitabine hydrochloride.
* Correlate EuroQOL ratings with those using symptom instruments (MSAS-SF) and quality of life instruments (FACT-G).
* Evaluate changes in perceived QOL, as measured by the EuroQOL instrument, and how these changes relate to symptom response and QOL response.
* Evaluate the patient's assessment of treatment burden, as measured by a single question, and how this compares to symptom response and QOL response.

OUTLINE: This is an open-label, multicenter study.

Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43, followed by 1 week of rest (course 1). For all subsequent courses, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life (QOL) and symptom response are assessed at baseline and at weeks 8, 16, and 32 (end of treatment). Questionnaires include the Memorial Symptom Assessment Scale-Short Form, Functional Assessment of Cancer Therapy-General, Pain Visual Analog Scale, and EuroQOL. Patients' perception of symptom response and perception of treatment burden are also assessed.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 52 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed poorly differentiated carcinoma or adenocarcinoma of unknown primary

  * Diagnosis based on biopsy and conventional imaging, including CT scans of the chest, abdomen, and pelvis with or without positron emission tomography (PET) scans or other specialized tests, performed within the past 4 weeks
* Must not have any of the following clinical features:

  * Squamous cell carcinoma in the lymph nodes of the neck or inguinal nodes only
  * Women with axillary lymph node metastases only
  * Women with peritoneal carcinomatosis only
  * Well-differentiated neuroendocrine tumors
  * Poorly differentiated tumors with midline tumor or elevated human chorionic gonadotropin (HCG)/alpha-fetoprotein (AFP)
  * Men with adenocarcinoma and elevated prostate-specific antigen (PSA)
* Measurable disease
* No symptom emergency at the time of study entry including, but not limited to, the following:

  * Back pain with epidural cord compression
  * Large effusions causing distress
  * Hypercalcemia
  * Bowel obstruction
  * Very painful (worst pain 10/10) solitary bone metastases with impending fracture

PATIENT CHARACTERISTICS:

* Modified "Physical Well-Being" subscale of the FACT-G score ≥ 6 within the past week
* Pain-intensity score ≥ 20 mm on the Memorial Pain Assessment Card OR receiving analgesics of ≥ 10 mg per day of oral morphine equivalent within the past week
* ECOG performance status 1-2
* WBC ≥ 3,000/mm³
* Platelet count ≥ 100,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to read, understand, and complete the quality of life and symptom questionnaires, and perception of change
* Able to complete the analgesic diary on a daily basis

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiation therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Efficacy, in terms of improved quality of life and reduction of symptom distress

SECONDARY OUTCOMES:
Changes in symptom distress, pain, and quality of life at 8, 16, and 32 weeks
Tumor response and duration
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Victor T. Chang, MD, Study Chair — Veterans Affairs Medical Center - East Orange; Raymond S. Lord, MD — West Michigan Cancer Center
Locations (37):
- United States (37):
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin